CLINICAL TRIAL: NCT02439320
Title: A Study of Two Doses of LAsMiditan (100 mg and 200 mg) Compared to Placebo in the AcUte Treatment of MigRAIne: A Randomized, Double-blind, Placebo-controlled Parallel Group Study
Brief Title: Lasmiditan Compared to Placebo in the Acute Treatment of Migraine:
Acronym: SAMURAI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16888; H8H-CD-LAHJ (Other: Eli Lilly and Company); COL MIG-301 (Other: CoLucid Pharmaceuticals)
Record Dates: First submitted 2015-03-18; First posted 2015-05-08 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Acute Migraine
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lasmiditan 100 mg (Experimental): Oral tablet. Lasmiditan 100 mg plus placebo (to match 200 mg tablet). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed within 24 hours.
  Interventions: Drug: Lasmiditan 100 mg; Drug: Placebo (matches lasmiditan doses)
- Lasmiditan 200 mg (Experimental): Oral tablet. Lasmiditan 200 mg plus placebo (to match 100 mg tablet). One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed within 24 hours.
  Interventions: Drug: Lasmiditan 200 mg; Drug: Placebo (matches lasmiditan doses)
- Placebo (Placebo Comparator): Oral tablet. Placebo tablets match lasmiditan 100 mg and lasmiditan 200 mg. One dose for acute treatment of migraine. Second dose for rescue or recurrence of migraine allowed within 24 hours.
  Interventions: Drug: Placebo (matches lasmiditan doses)

INTERVENTIONS:
Drug: Lasmiditan 100 mg
  Other Names: LY573144
  Arms: Lasmiditan 100 mg
Drug: Lasmiditan 200 mg
  Other Names: LY573144
  Arms: Lasmiditan 200 mg
Drug: Placebo (matches lasmiditan doses)

SUMMARY:
This is a prospective randomized, double-blind, placebo-controlled study in participants with disabling migraine (Migraine Disability Assessment (MIDAS) score ≥ 11).

DETAILED DESCRIPTION:
Participants will be asked to treat a migraine attack with study drug on an outpatient basis. Participants will be provided with a dosing card containing a dose for initial treatment and a second dose to be used for rescue or recurrence of migraine. Each participant's study participation will consist of a screening visit (Visit 1) with a telephone contact within 7 days to confirm eligibility, a Treatment Period of up to 8 weeks, and an End-of-Study (EoS) visit (Visit 2) within one week (7 days) of treating a single migraine attack. The total time on study is approximately 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Participants with migraine with or without aura fulfilling the International Headache Society (IHS) diagnostic criteria 1.1 and 1.2.1 (International Headache Classification (ICHD) 2004).
* History of disabling migraine for at least 1 year.
* MIDAS score ≥11.
* Migraine onset before the age of 50 years.
* History of 3 - 8 migraine attacks per month (< 15 headache days per month).
* Male or female, aged 18 years or above.
* Females of child-bearing potential must be using or willing to use a highly effective form of contraception (e.g. combined oral contraceptive, intrauterine device (IUD), abstinence or vasectomized partner).
* Able and willing to complete an electronic diary.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Known coronary artery disease, clinically significant arrhythmia or uncontrolled hypertension.
* History or evidence of hemorrhagic stroke, epilepsy or any other condition placing the participant at increased risk of seizures.
* History of recurrent dizziness and/or vertigo including benign paroxysmal positional vertigo (BPPV), Meniere's disease, vestibular migraine, and other vestibular disorders.
* History of diabetes mellitus with complications (diabetic retinopathy, nephropathy or neuropathy).
* History within the previous three years or current evidence of abuse of any drug, prescription or illicit, or alcohol.
* History of orthostatic hypotension with syncope.
* Significant renal or hepatic impairment.
* Participant is at imminent risk of suicide (positive response to question 4 or 5 on the C-SSRS) or had a suicide attempt within six months prior to the screening visit.
* Known Hepatitis B or C or HIV infection.
* History, within past 12 months, of chronic migraine or other forms of primary or secondary chronic headache disorder (e.g. hemicranias continua, medication overuse headache) where headache frequency is greater than 15 headache days per month.
* Use of more than 3 doses per month of either opiates or barbiturates.
* Initiation of or a change in concomitant medication to reduce the frequency of migraine episodes within three (3) months prior to Screening/Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2231 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (90):
- United States (90):
  - Southview Medical Group, P.C., Birmingham, Alabama
  - Simon-Williamson Clinic, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - East Valley Family Physicians, PC, Chandler, Arizona
  - Radiant Research,Inc, Chandler, Arizona
  - Warner Family Practice, Chandler, Arizona
  - Clinical Research Advantage/Fountain Hills Family Practice, Fountain Hills, Arizona
  - Neurological Physicians of Arizona, Inc, Gilbert, Arizona
  - Thunderbird Internal Medicine, Glendale, Arizona
  - Lenzmeier Family Practice, Glendale, Arizona
  - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Family Practice Specialists, Ltd, Phoenix, Arizona
  - Clinical Research Advantage Inc./Central Phoenix Medical Center LLC, Phoenix, Arizona
  - Thunderbird Internal Medicine, Phoenix, Arizona
  - Tatum Highlands Medical Associates, PLLC, Phoenix, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Arizona Community Physicians, Tucson, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Cassidy Medical Group, Carlsbad, California
  - Allied Clinical Research, Gold River, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - Cassidy Medical Group, Vista, California
  - Mile High Primary Care, Aurora, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - Clinical Research Advantage Inc/Colorado Springs Family Practice, Colorado Springs, Colorado
  - Comprehensive Clinical Development- Washington DC, Washington D.C., District of Columbia
  - Meridien Research, Brooksville, Florida
  - MD Clinical, Hallandale, Florida
  - Suncoast Research Group, Miami, Florida
  - CNS Healthcare, Orlando, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Meridien Research, Tampa, Florida
  - Radiant Research Inc, Atlanta, Georgia
  - Urban Family Practice, Marietta, Georgia
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Michigan Avenue Internists, Chicago, Illinois
  - Medical and Procedural Specialists of Illinois, Chicago, Illinois
  - Radiant Research, Inc, Chicago, Illinois
  - Evanston Premier Research LLC, Evanston, Illinois
  - Clinical Research Advantage, Evansville, Indiana
  - Family Medical Associates, Evansville, Indiana
  - Ridge Family Practice, Council Bluffs, Iowa
  - Radiant Research Inc./Continuum Health Care, Overland Park, Kansas
  - Heartland Research, Wichita, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - Radiant Research, Inc, Edina, Minnesota
  - West Florissant Internists, Bridgeton, Missouri
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, Inc, St Louis, Missouri
  - Skyline Medical Center, Elkhorn, Nebraska
  - Prairie Fields Family Medicine PC, Fremont, Nebraska
  - Southwest Family Physicians, PC, Omaha, Nebraska
  - James Mell, DO, Henderson, Nevada
  - Clinical Research Advantage, Henderson, Nevada
  - Nevada Family Care, Henderson, Nevada
  - Diagnostic Center of Medicine, Las Vegas, Nevada
  - Clifford Molin/Clinical Research Advantage,Inc, Las Vegas, Nevada
  - Comprehensive Clinical Development - Queens NY, Jamaica, New York
  - Radiant Research,Inc, Akron, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Radiant Research, Inc, Columbus, Ohio
  - Oklahoma City Clinic - Edmund, Edmond, Oklahoma
  - Oklahoma City Clinic - Midwest CIty, Midwest City, Oklahoma
  - LION Research, Norman, Oklahoma
  - Oklahoma City Clinic- Central/Clinical Research Advantage INC, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sunstone Medical Research,LLC, Medford, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Bay Clinical Research, Warwick, Rhode Island
  - Primary Care Associates, PA, Anderson, South Carolina
  - Radiant Research, Inc, Anderson, South Carolina
  - Medical Research South, Charleston, South Carolina
  - Radiant Research, Inc, Greer, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Family Medical Associates of Texas, Allen, Texas
  - Premier Family Physicians, Austin, Texas
  - Radiant Research, Inc, Dallas, Texas
  - Village Health Center, Plano, Texas
  - Doctors of Internal Medicine, Plano, Texas
  - Plano Internal Medicine, Plano, Texas
  - Radiant Research, San Antonio, Texas
  - Radiant Research, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Johnston KM, Powell L, Popoff E, Harris L, Croop R, Coric V, L'Italien G. Rimegepant, Ubrogepant, and Lasmiditan in the Acute Treatment of Migraine Examining the Benefit-Risk Profile Using Number Needed to Treat/Harm. Clin J Pain. 2022 Nov 1;38(11):680-685. doi: 10.1097/AJP.0000000000001072. PMID 36125279
- [Derived] Doty EG, Hauck PM, Krege JH, Komori M, Hake AM, Dong Y, Lipton RB. The Association Between the Occurrence of Common Treatment-Emergent Adverse Events and Efficacy Outcomes After Lasmiditan Treatment of a Single Migraine Attack: Secondary Analyses from Four Pooled Randomized Clinical Trials. CNS Drugs. 2022 Jul;36(7):771-783. doi: 10.1007/s40263-022-00928-y. Epub 2022 Jul 2. PMID 35779194
- [Derived] Krege JH, Lipton RB, Baygani SK, Komori M, Ryan SM, Vincent M. Lasmiditan for Patients with Migraine and Contraindications to Triptans: A Post Hoc Analysis. Pain Ther. 2022 Jun;11(2):701-712. doi: 10.1007/s40122-022-00388-8. Epub 2022 Apr 26. PMID 35471625
- [Derived] Charleston L 4th, Savage-Edwards B, Bragg SM, Baygani SK, Dennehy EB. Migraine history and response to lasmiditan across racial and ethnic groups. Curr Med Res Opin. 2022 May;38(5):721-730. doi: 10.1080/03007995.2022.2057152. Epub 2022 Apr 3. PMID 35350937
- [Derived] Reuter U, Krege JH, Lombard L, Gomez Valderas E, Krikke-Workel J, Dell-Agnello G, Dowsett SA, Buse DC. Lasmiditan efficacy in the acute treatment of migraine was independent of prior response to triptans: Findings from the CENTURION study. Cephalalgia. 2022 Jan;42(1):20-30. doi: 10.1177/03331024211048507. Epub 2021 Oct 13. PMID 34644189
- [Derived] Lipton RB, Baygani SK, Tepper SJ, Krege JH, Vasudeva R, Pearlman EM, Hauck PM, Loo LS. A close association of freedom from pain, migraine-related functional disability, and other outcomes: results of a post hoc analysis of randomized lasmiditan studies SAMURAI and SPARTAN. J Headache Pain. 2021 Aug 28;22(1):101. doi: 10.1186/s10194-021-01303-w. PMID 34454420
- [Derived] Martin VT, Ahmed Z, Hochstetler HM, Baygani SK, Dong Y, Hauck PM, Khanna R. Tolerability and Safety of Lasmiditan Treatment in Elderly Patients With Migraine: Post Hoc Analyses From Randomized Studies. Clin Ther. 2021 Jun;43(6):1066-1078. doi: 10.1016/j.clinthera.2021.04.004. Epub 2021 Aug 6. PMID 34366152
- [Derived] Peres MFP, Vasudeva R, Baygani SK, Dennehy EB, Vincent M, Friedman DI. Lasmiditan efficacy in migraine attacks with mild vs. moderate or severe pain. Curr Med Res Opin. 2021 Jun;37(6):1031-1038. doi: 10.1080/03007995.2021.1903846. Epub 2021 Apr 7. PMID 33784930
- [Derived] Clemow DB, Hochstetler HM, Dong Y, Hauck P, Peres MFP, Ailani J. Effect of a change in lasmiditan dose on efficacy and safety in patients with migraine. Postgrad Med. 2021 May;133(4):449-459. doi: 10.1080/00325481.2020.1860619. Epub 2021 Mar 17. PMID 33730977
- [Derived] Clemow DB, Baygani SK, Hauck PM, Hultman CB. Lasmiditan in patients with common migraine comorbidities: a post hoc efficacy and safety analysis of two phase 3 randomized clinical trials. Curr Med Res Opin. 2020 Nov;36(11):1791-1806. doi: 10.1080/03007995.2020.1808780. Epub 2020 Oct 6. PMID 32783644
- [Derived] Smith T, Krege JH, Rathmann SS, Dowsett SA, Hake A, Nery ESM, Matthews BR, Doty EG. Improvement in Function after Lasmiditan Treatment: Post Hoc Analysis of Data from Phase 3 Studies. Neurol Ther. 2020 Dec;9(2):459-471. doi: 10.1007/s40120-020-00185-5. Epub 2020 May 23. PMID 32447545
- [Derived] Knievel K, Buchanan AS, Lombard L, Baygani S, Raskin J, Krege JH, Loo LS, Komori M, Tobin J. Lasmiditan for the acute treatment of migraine: Subgroup analyses by prior response to triptans. Cephalalgia. 2020 Jan;40(1):19-27. doi: 10.1177/0333102419889350. Epub 2019 Nov 19. PMID 31744319
- [Derived] Ashina M, Vasudeva R, Jin L, Lombard L, Gray E, Doty EG, Yunes-Medina L, Kinchen KS, Tassorelli C. Onset of Efficacy Following Oral Treatment With Lasmiditan for the Acute Treatment of Migraine: Integrated Results From 2 Randomized Double-Blind Placebo-Controlled Phase 3 Clinical Studies. Headache. 2019 Nov;59(10):1788-1801. doi: 10.1111/head.13636. Epub 2019 Sep 17. PMID 31529622
- [Derived] Shapiro RE, Hochstetler HM, Dennehy EB, Khanna R, Doty EG, Berg PH, Starling AJ. Lasmiditan for acute treatment of migraine in patients with cardiovascular risk factors: post-hoc analysis of pooled results from 2 randomized, double-blind, placebo-controlled, phase 3 trials. J Headache Pain. 2019 Aug 29;20(1):90. doi: 10.1186/s10194-019-1044-6. PMID 31464581
- [Derived] Loo LS, Plato BM, Turner IM, Case MG, Raskin J, Dowsett SA, Krege JH. Effect of a rescue or recurrence dose of lasmiditan on efficacy and safety in the acute treatment of migraine: findings from the phase 3 trials (SAMURAI and SPARTAN). BMC Neurol. 2019 Aug 13;19(1):191. doi: 10.1186/s12883-019-1420-5. PMID 31409292
- [Derived] Loo LS, Ailani J, Schim J, Baygani S, Hundemer HP, Port M, Krege JH. Efficacy and safety of lasmiditan in patients using concomitant migraine preventive medications: findings from SAMURAI and SPARTAN, two randomized phase 3 trials. J Headache Pain. 2019 Jul 24;20(1):84. doi: 10.1186/s10194-019-1032-x. PMID 31340760
- [Derived] Doty EG, Krege JH, Jin L, Raskin J, Halker Singh RB, Kalidas K. Sustained responses to lasmiditan: Results from post-hoc analyses of two Phase 3 randomized clinical trials for acute treatment of migraine. Cephalalgia. 2019 Oct;39(12):1569-1576. doi: 10.1177/0333102419859313. Epub 2019 Jul 3. PMID 31266353
- [Derived] Krege JH, Rizzoli PB, Liffick E, Doty EG, Dowsett SA, Wang J, Buchanan AS. Safety findings from Phase 3 lasmiditan studies for acute treatment of migraine: Results from SAMURAI and SPARTAN. Cephalalgia. 2019 Jul;39(8):957-966. doi: 10.1177/0333102419855080. Epub 2019 Jun 5. PMID 31166697
- [Derived] Tepper SJ, Krege JH, Lombard L, Asafu-Adjei JK, Dowsett SA, Raskin J, Buchanan AS, Friedman DI. Characterization of Dizziness After Lasmiditan Usage: Findings From the SAMURAI and SPARTAN Acute Migraine Treatment Randomized Trials. Headache. 2019 Jul;59(7):1052-1062. doi: 10.1111/head.13544. Epub 2019 Jun 1. PMID 31152441
- [Derived] Kuca B, Silberstein SD, Wietecha L, Berg PH, Dozier G, Lipton RB; COL MIG-301 Study Group. Lasmiditan is an effective acute treatment for migraine: A phase 3 randomized study. Neurology. 2018 Dec 11;91(24):e2222-e2232. doi: 10.1212/WNL.0000000000006641. Epub 2018 Nov 16. PMID 30446595

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a double-blind, placebo-controlled parallel group study.
Groups:
- 100 mg Lasmiditan: 100 milligrams (mg) lasmiditan administered PO within 4 hours of onset of migraine attack. If the migraine did not respond 2 hours postdose a second dose of study drug can be taken up to 24 hours after the first dose.
- 200 mg Lasmiditan: 200 milligrams (mg) lasmiditan administered PO within 4 hours of onset of migraine attack. If the migraine did not respond 2 hours postdose a second dose of study drug can be taken up to 24 hours after the first dose.
- Placebo: Placebo administered PO within 4 hours of onset of migraine attack. If the migraine did not respond 2 hours postdose a second dose of study drug can be taken up to 24 hours after the first dose.
Period: Overall Study
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Started | 744 | 745 | 742
Confirmed Eligibility | 710 | 695 | 705
1st Dose (by 4 Hours Migraine Onset) (Safety population based on the first dose. Participants received at least 1 dose of study drug.) | 630 | 609 | 617
2nd Dose (After 2 Hour Assessment) (Participants received second dose of study drug after 4 hours.) | 289 | 238 | 401
Completed (Included participants who received study drug and participants who did not receive study drug.) | 648 | 631 | 643
Not Completed | 96 | 114 | 99
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 37 | 34 | 42
Not completed — Death | 0 | 1 | 0
Not completed — Noncompliance with Protocol | 10 | 11 | 7
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 12 | 16 | 14
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Sponsor Request | 0 | 2 | 1
Not completed — Randomization Failure | 35 | 46 | 34

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo | Total
Number analyzed (Participants) | 630 | 609 | 617 | 1856
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.67) | 41.4 (12.04) | 42.4 (12.30) | 42.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 512 | 515 | 525 | 1552
  Male | 118 | 94 | 92 | 304
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 82 | 77 | 84 | 243
  Not Hispanic or Latino | 544 | 527 | 529 | 1600
  Unknown or Not Reported | 4 | 5 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unknown or Not reported row is listed as Other in the Clinical Study Report.
  Participants
    American Indian or Alaska Native | 7 | 7 | 1 | 15
    Asian | 4 | 4 | 2 | 10
    Native Hawaiian or Other Pacific Islander | 1 | 3 | 2 | 6
    Black or African American | 122 | 125 | 119 | 366
    White | 471 | 450 | 479 | 1400
    More than one race | 11 | 6 | 6 | 23
    Unknown or Not Reported | 14 | 14 | 8 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 630 | 609 | 617 | 1856
Duration of Migraine History [Mean (Standard Deviation); unit: years] | 19.7 (12.98) | 18.9 (13.12) | 19.3 (12.65) | 19.3 (12.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Headache Pain Free
Description: The percentage of participants defined as mild, moderate, or severe headache pain becoming none.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable headache pain free data.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 503 | 518 | 524
percentage of participants | 28.2 | 32.2 | 15.3
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.6 to 3.0]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.6, 95% CI 2-sided [2.0 to 3.6]

2. Primary Outcome: Percentage of Participants Who Are Most Bothersome Symptom (MBS) Free
Description: The percentage of participants defined as the associated symptom present and identified as MBS (nausea, photophobia, or phonophobia) prior to dosing being absent.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable MBS data.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 469 | 481 | 488
percentage of participants | 40.9 | 40.7 | 29.5
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.3 to 2.2]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 1.6, 95% CI 2-sided [1.3 to 2.1]

3. Secondary Outcome: Percentage of Participants Who Have Headache Relief After First Dose
Description: The percentage of participants with headache pain moderate or severe which became mild or none or with headache pain mild which became none.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable headache relief data.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 59.4 | 59.5 | 42.2
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 2.4, 95% CI 2-sided [1.8 to 3.1]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.9 to 3.3]

4. Secondary Outcome: Percentage of Participants With Headache Recurrence
Description: Participants who received study drug and which became pain free at 2 hours post-dose and worsened again up to 48 hours post-dose.
Time Frame: From 2 hours post dose up to 48 hours
Population: Randomized participants who received a dose of study drug and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 8.4 | 10.1 | 5.1
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.1 to 2.8]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.3 to 3.4]

5. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: Rescue medication was permitted after completion of the 2 hour assessment if the migraine did not respond (participant was not pain free).
Time Frame: 2 hours post dose
Population: Randomized participants who received a dose of study drug and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 26.2 | 20.7 | 46.0
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.3 to 0.5]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.3, 95% CI 2-sided [0.2 to 0.4]

6. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: as for outcome 5
Time Frame: Anytime between 2-24 hours post dose
Population: Randomized participants who received a dose of study drug and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 255
percentage of participants | 8.9 | 7.9 | 11.7
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.120, Regression, Logistic; Odds Ratio, log = 0.7, 95% CI 2-sided [0.5 to 1.1]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.035, Regression, Logistic; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.4 to 1.0]

7. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: as for outcome 5
Time Frame: Anytime 24-48 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable use of rescue medication data.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Nausea Free
Description: The percentage of participants without nausea.
Time Frame: 2 hours post dose
Population: All randomized participants who used at least 1 dose of study drug and had any post-dose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 64.6 | 64.1 | 62.1
Statistical Analysis 1: Comparison: 100 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.386, Regression, Linear; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.9 to 1.4]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan vs Placebo; Test type: Superiority; p = 0.470, Regression, Linear; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.9 to 1.4]

9. Secondary Outcome: Percentage of Participants Phonophobia Free
Description: The percentage of participants without phonophobia.
Time Frame: 2 hours post dose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 60.7 | 58.7 | 52.5
Statistical Analysis 1: Comparison: 100 mg Lasmiditan; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.1 to 1.8]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI 2-sided [1.0 to 1.6]

10. Secondary Outcome: Percentage of Participants Photophobia Free
Description: The percentage of participants without photophobia.
Time Frame: 2 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable photophobia free data.
Measure: Number; unit: percentage of participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 562 | 555 | 554
percentage of participants | 53.9 | 51.5 | 38.1
Statistical Analysis 1: Comparison: 100 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.5 to 2.4]
Statistical Analysis 2: Comparison: 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.4 to 02.2]

11. Secondary Outcome: Participants With Serious Adverse Events (SAE)
Description: Safety and Tolerability was assessed by the number of participants with at least 1 treatment emergent event (TEAE). A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section
Time Frame: Baseline up to 11 weeks
Population: All randomized participants who had received at least one dose of study drug. Results are displayed by the first dose taken.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
Number analyzed (Participants) | 630 | 609 | 617
Participants | 0 | 2 | 1

12. Other Pre Specified Outcome: Percentage of Participants With Resource Utilization
Description: Use of health care for treatment 6 months prior to enrolling in the study and information reported during time on study
Time Frame: 6 months prior to enrolling in study to end of study (Up to 11 Weeks) within 7 days of treating a single migraine attack
Population: All randomized participants who used at least 1 dose of study drug, regardless of whether or not they underwent any study assessments.
Measure: Number; unit: percentage of participants
Groups:
- 100 mg Lasmiditan/100 mg Lasmiditan; 200 mg Lasmiditan/200 mg Lasmiditan: 100 milligrams (mg) lasmiditan administered PO within 4 hours of onset of migraine attack. An optional 100 mg Lasmiditan dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- 100 mg Lasmiditan/Placebo: 100 milligrams (mg) lasmiditan administered PO within 4 hours of onset of migraine attack. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- 200 mg Lasmiditan/Placebo: 200 milligrams (mg) lasmiditan administered PO within 4 hours of onset of migraine attack. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
- Placebo/Placebo: Placebo tablets match each of the lasmiditan doses (100 mg and 200 mg) was administered orally, once for acute treatment of migraine. A second optional dose was administered between 2 and 24 hours for rescue or recurrence of migraine.
Arm/Group | 100 mg Lasmiditan/100 mg Lasmiditan | 100 mg Lasmiditan/Placebo | 200 mg Lasmiditan/200 mg Lasmiditan | 200 mg Lasmiditan/Placebo | Placebo/Placebo
Number analyzed (Participants) | 433 | 197 | 406 | 203 | 617
percentage of participants
  6 Months prior to enrolling | 4.4 | 4.6 | 3.0 | 2.5 | 2.8
  During time of study | 0.9 | 0.5 | 0.2 | 0.5 | 0.6

ADVERSE EVENTS:
Time Frame: up to 11 weeks
Description: All randomized participants who had received at least one dose of study drug.
Groups:
- 100 mg Lasmiditan: Any participant who received 100 milligrams (mg) lasmiditan administered PO.
- 200 mg Lasmiditan: Any participant who received 200 milligrams (mg) lasmiditan administered PO.
- Placebo: Any participant who received placebo administered PO.
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/630 | 0/609 | 0/617
Serious Adverse Events (participants affected / at risk) | 0/630 | 2/609 | 1/617
Other Adverse Events (participants affected / at risk) | 258/630 | 280/609 | 113/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Lasmiditan (N=630) | 200 mg Lasmiditan (N=609) | Placebo (N=617)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 100 mg Lasmiditan (N=630) | 200 mg Lasmiditan (N=609) | Placebo (N=617)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 2 (2) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 6 (6) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (19) | 33 (33) | 14 (16)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7) | 5 (5)
Abasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 6 (6) | 7 (7) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 2 (2) | 3 (3)
Fatigue (General disorders) | 28 (28) | 21 (21) | 3 (3)
Feeling abnormal (General disorders) | 7 (7) | 4 (4) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 1 (1) | 1 (1)
Feeling drunk (General disorders) | 1 (1) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 1 (1)
Feeling jittery (General disorders) | 3 (3) | 3 (3) | 1 (1)
Feeling of relaxation (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (11) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 6 (6) | 7 (7) | 0 (0)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 87 (91) | 107 (114) | 22 (23)
Dysarthria (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 9 (10) | 12 (13) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 15 (16) | 17 (18) | 3 (3)
Mental impairment (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 42 (43) | 50 (51) | 14 (14)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Sedation (Nervous system disorders) | 3 (3) | 8 (8) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory integrative dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 40 (40) | 36 (37) | 14 (14)
Tremor (Nervous system disorders) | 7 (7) | 4 (4) | 1 (1)
Tunnel vision (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 5 (5) | 1 (1)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Blunted affect (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Depersonalisation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hypnagogic hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Listless (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Phonophobia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/525 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/525 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 5 (5) | 2 (2)
Hot flush (Vascular disorders) | 5 (5) | 3 (3) | 3 (3)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days